CLINICAL TRIAL: NCT06906159
Title: Cricket Protein Bioavailability in Younger, Middle-Aged and Alder Adults
Brief Title: Cricket Protein Bioavailability in Younger, Middle-Aged and Older Adults
Acronym: CriProB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: HOP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CriProB
Record Dates: First submitted 2025-01-08; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cricket Protein; Whey Protein
MeSH Terms: interventions — capsid protein, Cricket paralysis virus; Whey Proteins

STUDY DESIGN:
Intervention Model Description: Repeated measures randomised crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One member of the research team is in charge if blinding the muffins to 'A' and 'B'
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cricket muffin (Experimental): Muffin made with cricket-derived protein powder
  Interventions: Dietary Supplement: Cricket protein
- Whey muffin (Active Comparator): Muffin made with whey protein powder
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Cricket protein — Muffins made with cricket-derived protein from house crickets (Acheta domesticus )
  Arms: Cricket muffin
Dietary Supplement: Whey protein — Muffins made with whey protein
  Arms: Whey muffin

SUMMARY:
A global shift towards sustainable food sources is now emerging, largely due to the immense environmental pressure that comes from producing animal foods, particularly beef. Insects present a novel source of sustainable dietary protein due to their high protein content. This is particularly relevant for older adults, as protein becomes increasingly more important in later life. It helps to maintain muscle as we age, which is crucial for reducing frailty, falls and early mortality. We want to find out more about the digestion and absorption of insect protein in older people to see if it could be a beneficial source of protein to help maintain muscle. We are interested in the use of insect-based solid foods, especially the use of flour made from grounded whole crickets. We want to explore the digestibility of cricket protein compared to a commonly used animal alternative (whey protein) to find out if it can be efficiently absorbed and utilised within humans.

DETAILED DESCRIPTION:
Participants are asked to fast overnight and come in the following day for one of two visits where they are given a standardised breakfast muffin containing either cricket protein or whey protein (250-300 kcal; approx. 12% fat, 45% carbohydrates including 10% sugars, 35% protein, 0.4% salt and 6% fibre) after which they breathe into a test tube in 15-30 minute intervals for 4 hours. In addition to this, we collect a blood sample (10ml) every 15 minutes for the first hour and then every 30 minutes for the next 3 hours (110ml of blood in total per visit) so we can determine changes in blood amino acids, glucose and fat concentrations after eating the muffin. In total we only collect a small amount of blood. This method of blood collection is the same method used for a traditional blood test but to avoid repeated needle insertions we use a cannula which remains in the participant's arm for the duration of the visit so that only a single needle insertion is necessary.

The muffin contains a small amount of a natural fat called octanoic acid. The octanoic acid is enriched with carbon-13. This is a natural variant of carbon and is safe to use, even in babies and pregnant women. At the end of each test visit we ask participants to fill out a short questionnaire to ask about the taste of the muffins. Participants are required to repeat this whole process for a second visit in which they consume the other muffin.

The muffins are identical between the two test visits with the exception that one muffin is made with a milk-based protein (whey) whereas the other test muffin is made with an insect protein (cricket). The test muffins are similar in size, shape, and taste. Participants are randomised to a muffin condition in a crossover design. Participants are blinded to the muffin condition and only one member of the research team knows which muffin participants receive on which test visit but they are not present during the test visits. The researchers conducting the test visits do not know which muffin is being consumed by participants.

Participants are required to attend for 2 test visits each lasting approximately 5 hours. This takes place in the Clinical Investigation Unit (CIU) at the University of Surrey. On the day before each of the test visits participants are asked to arrive fasted for 12 hours overnight, refrain from strenuous exercise, alcohol, caffeine and food containing corn, broccoli, sugarcane, and tropical fruits (because of the type of natural carbon-13 they contain) the day before their visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females in general good health, aged between 18 - 35 years, 40 - 55 years or over 65 years
* BMI between 18.5 and 35 kg/m2
* Stable weight for at least 3 months
* Volunteers must be able and willing to give informed written consent
* Volunteers must be able to eat egg
* Volunteers must be willing to provide blood samples

Exclusion Criteria:

* Current or previous gastrointestinal conditions (e.g. Crohn's disease, Coeliac disease, Irritable Bowel Syndrome) - assessed via a health questionnaire
* Those with diabetes or other metabolic conditions - assessed via a health questionnaire
* Those taking food supplements which may impact digestion (e.g., digestive enzymes, probiotics, fibre supplements)
* Those smoking, using nicotine products (e.g., e-cigarettes, patches) or not abstained from these activities for more than 6 months - assessed via a health questionnaire
* Pregnant or lactating
* Volunteers with a high daily caffeine intake > 300 mg/day (more than 5 cups of standard coffee per day)
* Drug or alcohol abuse in the last 2 years
* Those who are currently taking part in a clinical trial or another research study or have taken part within the last 3 months
* Those with food allergies, dietary intolerance or Coeliac disease - assessed via a health questionnaire
* Those following weight loss diets

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | 4 hour post-prandial period
  Exhaled breath is used to assess the rate of gastric emptying of the protein muffins
Plasma amino acids | 4 hour post-prandial period
  Blood samples are used to assess the plasma amino acid response to consuming the protein muffins

SECONDARY OUTCOMES:
Metabolic markers | 4 hour post-prandial period
  Blood samples are also used to assess post-prandial glucose, triglycerides and cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: James Rutherford, MSc, Study Director — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No